CLINICAL TRIAL: NCT01118793
Title: PREDICT: Scripps Pilot Study on the Effect of High Clopidogrel Maintenance Dosing and Its Relationship to Cytochrome P450 2C19 Polymorphism Status
Brief Title: Pilot Study on the Effect of High Clopidogrel Maintenance Dosing
Acronym: PREDICT
Status: Completed | Type: Observational
Sponsor: Scripps Health (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: HSC# 08-5083; 1UL1RR025774-01 (NIH)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- double dosing of Clopidogrel: This is a Scripps pilot study on the effect of high clopidogrel maintenance dosing and its relationship to cytochrome P450 2C19 polymorphism status [STSI/CTSA].
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — 150 mg dosage of Clopidogrel for 7 to 10 days.
  Other Names: Plavix

SUMMARY:
This is a Scripps pilot study on the effect of high clopidogrel maintenance dosing and its relationship to cytochrome P450 2C19 polymorphism status [STSI/CTSA].

DETAILED DESCRIPTION:
When added to aspirin, clopidogrel at a routine dose of 75 mg daily reduces the incidence of thrombotic vascular adverse events in patients with acute coronary syndromes and those undergoing percutaneous interventions (PCI). The observation that many patients have less than expected platelet inhibition with clopidogrel has given rise to the concept of clopidogrel resistance. Clopidogrel resistance is associated with increased adverse events such as stent thrombosis, post-stent ischemic events and periprocedural myocardial infarctions. Some patients can overcome the resistance with increasing the dose of clopidogrel. A higher maintenance dose (150 mg daily) in patients undergoing PCI results in superior platelet inhibition and may reduce cardiovascular events. Clopidogrel is a thienopyridine prodrug, which is converted to its active metabolite by several enzymes of the P450 family, including CYP2C19. The loss-of-function CYP2C19*2 (681 G>A) single nucleotide polymorphism (SNP), occurring as either a hetero- or homozygous allele, reduces the conversion of clopidogrel to its active metabolite. Two recent studies have shown an association between CYP2C19*2 polymorphism and lack of platelet inhibition with clopidogrel. These studies included healthy volunteers and patients undergoing elective PCI and demonstrated a prevalence of the CYP2C19*2 allele of 25-30%. Platelet inhibition was not affected by clopidogrel in those who carried the CYP2C19*2 polymorphism.

Our hypothesis is the following: Patients who are carriers of the loss-of-function CYP2C19*2 allele (heterozygous 1*/2* or homozygous 2*/2*) have decreased platelet inhibition on clopidogrel which cannot be overcome with increasing the maintenance dose from 75 mg to 150 mg daily.

The specific aim will include an evaluation of the anti-platelet response of a higher maintenance dose of clopidogrel (150 mg /daily) in patients who are resistant to the usual dose (75 mg/daily) and are either carriers or non-carriers of the CYP2C19*2 allele.

The study design will be a single center, prospective, observational pilot study. We will screen and enroll patients who are followed at Scripps Clinic and on chronic clopidogrel therapy. All patients will be eligible. A blood sample will be collected to perform DNA extraction and genotyping for the CYP2C19*2 polymorphism. Platelet function assays will be performed using VerifyNow point-of-care assay. We will recruit 60 patients with high platelet reactivity (PRU > 230): 30 wild-types (normal) and 30 carriers (heterozygous or homozygous) of the CYP2C19*2 polymorphism. These patients will be given 150 mg of clopidogrel for 1 week, at which time the platelet assay will be repeated. At that time, patients will be counseled by the study physicians regarding the potential risks and benefits of continuing to receive 150 mg of clopidogrel per day versus returning to the FDA approved dose of 75 mg daily.

The immediate objective is to evaluate the possibility of overcoming clopidogrel resistance in carriers of CYP2C19*2 with a higher maintenance dose. The long term objective is to improve patient care and outcomes using personalized medicine based on the individual's genotype.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females between the ages of 18-85.
* Patients able to give informed written consent.
* Patients on clopidogrel for ≥ 7 days.

Exclusion Criteria:

* Participation in a study of experimental therapy or device within prior 30 days.
* Pregnant women or women of childbearing potential not using an acceptable method of contraception who have not been proven to have a negative pregnancy test result.
* Inability to comply with all aspects of the protocol.
* History of bleeding diathesis or evidence of active abnormal bleeding within previous 90 days.
* Severe hypertension (systolic blood pressure > 200 mm Hg or diastolic blood pressure > 110 mm Hg) not adequately controlled on antihypertensive therapy.
* Major surgery within the preceding 6 weeks.
* History of stroke within 30 days or any history of hemorrhagic stroke.
* History of intracranial neoplasm.
* Current or planned administration of another parenteral GP IIb-IIIa inhibitor within 7 days of enrollment.
* Known hypersensitivity to any component of the product.
* Unstable angina with dynamic ST or T wave changes within 48 hours of enrollment.
* Administration of LMWH within 8 hours prior to enrollment or UFH within 60 minutes unless a PPT < 50 secs or ACT < 150 secs.
* On chronic anticoagulation (i.e. Coumadin).
* Hemoglobin < 10 g/dL.
* Hematocrit < 30%.
* Platelet count < 100,000 mcL.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Scripps Health patients having decresed platlet inhibition on clopidogrel
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Barker, MD, Principal Investigator — Scripps Health
Locations (1):
- Scripp Health, La Jolla, California, United States